CLINICAL TRIAL: NCT06141785
Title: Early Nutritional Intervention to Prevent Malnutrition in Patients With Cancer Receiving Palliative Chemotherapy in an Outpatient Setting
Brief Title: Early Nutritional Intervention in Patients With Cancer
Acronym: NICOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Kirstine Guld Frederiksen, Principal investigator, Gødstrup Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGF-1-2023
Record Dates: First submitted 2023-11-07; First posted 2023-11-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Nutritional Intervention; Cancer; Malnutrition
Keywords: Nutritional interventions; Dietetics; Cancer; Malnutrition; Nutrition
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Intervention Model Description: Intervention with a historical control cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Intervention (Experimental): Patients with Cancer treated with palliative chemotherapy.
  Interventions: Other: Nutritional intervention
- Historical control (No Intervention): Patients with Cancer treated with palliative chemotherapy.
  Historical Control cohort following current clinical practise, where nutritional treatment is not systematically implemented but patients can be referred to a clinical dietitian after clinical assessment by the treating physician or nurse.

INTERVENTIONS:
Other: Nutritional intervention — An individually targeted nutritional intervention, and a simple home-based physical exercise program. The Nutritional intervention will be delivered by a clinical dietitian, from treatment initiation and throughout the treatment trajectory
  Arms: Nutritional Intervention

SUMMARY:
The goal of this intervention study is to study the effect of nutritional interventions in patients with cancer receiving palliative chemotherapy. The main question it aims to answer is: Does early nutritional interventions affect body weight, quality of life, survival, muscle mass, performance status, physical function, nutritional risk and treatment tolerance in patients with cancer receiving palliative chemotherapy? Researchers will compare patients receiving the intervention to a historical control cohort following current clinical practice.

DETAILED DESCRIPTION:
Background 30-50% of patients with cancer are malnourished, resulting in poorer prognosis, increased toxicities, reduced quality of life, and reduced physical function. Nevertheless, cancer-related malnutrition remains largely unrecognized and undertreated in clinical practice.

Aim To examine the effect of an early individualised nutritional intervention on body weight, quality of life, survival, muscle mass, performance status, physical function, nutritional risk, and treatment tolerance in patients with cancer receiving palliative chemotherapy.

Methods An intervention study with a historical control cohort. Participants are newly diagnosed patients with lung, pancreatic, ovarian, or colorectal cancers recruited at initiation of palliative chemotherapy. The control group followed current clinical practice. The intervention group receives an individualised nutritional intervention delivered by a clinical dietitian from treatment initiation and throughout the treatment trajectory. The intervention is tailored to the participant's nutritional needs, food preferences, nutrition impact symptoms, and smell- and taste disorders. The primary endpoint is change in body weight. Secondary endpoints include quality of life, survival, muscle mass, performance status, physical function, nutritional risk, and treatment tolerance. Data are collected at baseline and after 12 and 24 weeks.

Perspectives The project will provide new knowledge on the effects of individualised nutritional interventions for patients with cancer receiving palliative chemotherapy, and the potential to improve quality of life, treatment tolerance, and survival.

ELIGIBILITY:
Inclusion Criteria:

* patients who are newly diagnosed with lung, colorectal, ovarian, or pancreatic cancer.
* patients treated with first-line palliative chemotherapy
* patients who are Danish speaking
* patients ≥18 years of age
* patients who are cognitive well-functioning

Exclusion Criteria:

* Patients not using electronic mail
* patients with dementia
* patients not able to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Body weight | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  Change in body weight in kilogram

SECONDARY OUTCOMES:
Self reported Quality of life | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  Measured by the questionnaire European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group (QLG) Core Questionnaire: Quality of Life (QLQ) Core 30 (EORTC QLQ-C30) using a Likert scale ranging from 1 to 4 for questions regarding function and symptoms, where a high score corresponds to a worse outcome, and a Likert scale ranging from 1 to 7 for questions regarding Global Health Status and Quality of Life, where a high score corresponds to a better outcome.
Survival | one year after initiation
  one-year survival will be assessed in the electronic patient journal
Muscle mass | baseline and week 24 (±2 weeks)
  CT scans to measure paraspinal muscle mass at the level of lumbal spine 3 (L3) which will also be assessed using measurements from the bio impedance scale
Performance status | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  Patient's performance status will be assessed by the treating physician according to the Eastern Cooperative Oncology Group (ECOG) classification on a scale ranging from 0 to 5, where a high score corresponds to a worse outcome
Hand grip strength | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  The Hand grip strength as a measure of physical function will be estimated. Hand grip strength will be measured using a hand dynamometer ("CAMRY" Digital Hand Dynamometer). The hand grip strength will be measured three times in the dominant hand, and the highest value in kilogram is registered.
Timed up and go | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  Timed up and go, as a measure om physical function, will be performed in the hallway from a chair with armrest. The patient is asked to walk three meters to a marked spot on the floor, return and sit down as quickly as possible without running. The test is performed twice, and the quickest time measurement is registered. The result is registered in seconds.
Nutritional Risk | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  To assess the nutritional risk, the patient will be screened by Nutrition Risk Screening 2002 (NRS-2002). This tool calculates a score based on information about Body Mass Index, weight loss, nutritional intake, severity of disease, and age. Results can be between 0 and 7, where a high score corresponds to a worse outcome
Dose intensity | baseline, week 12 (±2 weeks), week 24 (±2 weeks)
  As a measure of treatment tolerance, dose intensity is registered on a scale ranging from 0 to -2, where 0 corresponds to a better outcome
Chemotherapy | week 12 (±2 weeks), week 24 (±2 weeks)
  As a measure of treatment tolerance, any change in chemotherapy drug will be registered
Duration of chemotherapy | week 24 (±2 weeks)
  As a measure of treatment tolerance, the duration of treatment with chemotherapy will be registered in days
Postponements in chemotherapy treatment | week 12 (±2 weeks), week 24 (±2 weeks)
  As a measure of treatment tolerance, the number of postponements of chemotherapy will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Ovesen, Prof, Study Director — University Clinic for Flavour, Balance and Sleep
Locations (1):
- Gødstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No